CLINICAL TRIAL: NCT03496077
Title: Addictive Potential of Little Cigars/Cigarillos in Dual Users: Effect by Flavor and Gender
Brief Title: Addictive Potential of LCCs in Dual Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Erin Mead-Morse, Assistant Professor, UConn Health
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 18-091-1
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Tobacco Use Disorder; Dual Tobacco Use; Tobacco Dependence; Smoking; Smoking, Cigar; Smoking, Cigarette; Smoking, Tobacco
Keywords: Dual Use; Little Cigars and Cigarillos; Cigarettes; Flavored Tobacco Use; Addiction Potential
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Cigar Smoking; Cigarette Smoking; Tobacco Smoking | interventions — Flavoring Agents; Tobacco Products

STUDY DESIGN:
Intervention Model Description: Randomized cross-over study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flavored LCCs (Experimental): Half of the group will start with a flavored little cigar/cigarillo (LCC) and cross over to unflavored LCC. The LCCs will be a popular brand already available for sale on the market.
  Interventions: Other: Flavored and unflavored little cigars/cigarillos (LCCs)
- Unflavored LCCs (Experimental): Half of the group will start with an unflavored little cigar/cigarillo (LCC) and cross over to flavored LCC. The LCCs will be a popular brand already available for sale on the market.
  Interventions: Other: Flavored and unflavored little cigars/cigarillos (LCCs)

INTERVENTIONS:
Other: Flavored and unflavored little cigars/cigarillos (LCCs) — Flavored and unflavored LCCs that are currently available for purchase

SUMMARY:
This study is about whether or not little cigars and cigarillos cause or maintain addiction, and if flavors, such as fruit, make them more addictive. The purpose of this study is to understand the addiction potential of little cigars and cigarillos compared to cigarettes in young adults who smoke both products. This study will also look at the differences between men and women. In the rest of this form, little cigars or cigarillos will be referred to as LCCs.

ELIGIBILITY:
Inclusion Criteria:

* Current regular dual user of little cigars/cigarillos (LCCs) and cigarettes, defined as: (a) report smoking cigarettes on ≥ 8 of the past 30 days, and (b) report smoking unaltered LCCs (without marijuana) on ≥ 8 of the past 30 days.
* Able to speak, read and understand English
* Age 18-34 years of age
* Stable residence (not planning to move during study period)
* Not intending to quit smoking cigarettes or LCCs within the next 2 weeks
* An expired carbon monoxide (CO) level of at least 4 ppm of expired air to verify smoking status

Exclusion Criteria:

* Pregnant for women (verified by urine pregnancy test at Visits 1 and 2)
* Current use of (or plans to use in the next 2-3 weeks) nicotine replacement products or cessation products (e.g., bupropion) to minimize confounding effects of another product)
* Positive breath alcohol screen (breath alcohol level (BAL) > 0 g/ml; one re-test allowed; assessed at Visits 1, 2, and 3)
* Illicit drug use other than marijuana (verified by positive drug toxicology test at Visits 1 and 3; one re-test allowed)
* Met criteria for Cannabis Dependence assessed by the Cannabis Use Disorders Identification Test-Revised (CUDIT-R)

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Demand elasticity for preferred flavor LCCs | Post-treatment (after being assigned to use it for 7 days)
  It is measured by the Cigarette Purchase Task, which will be adapted to assess this product. It is the hypothetical consumption of preferred flavor LCCs as increasing prices on a log-log scale.
Demand elasticity for unflavored LCCs | Post-treatment (after being assigned to use it for 7 days)
  It is measured by the Cigarette Purchase Task, which will be adapted to assess this product. It is the hypothetical consumption of unflavored LCCs as increasing prices on a log-log scale.

CONTACTS AND LOCATIONS:
Overall Officials: Erin L Mead, PhD,MHS, Principal Investigator — UConn Health, Farmington, CT
Locations (1):
- UConn Health, Farmington, Connecticut, United States